CLINICAL TRIAL: NCT05941754
Title: A Clinical Study of Omega-3 on Depression and Cognition
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NFEC-2023-051
Record Dates: First submitted 2023-02-15; First posted 2023-07-12 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Depression
Keywords: omega-3; cognition; depression
MeSH Terms: conditions — Depression | interventions — Docosahexaenoic Acids

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- high omega-3 group (Experimental): A single dose of 4.0g EPA was given orally
  Interventions: Dietary Supplement: omega-3
- low omega-3 group (Experimental): A single dose of 2.0g EPA was given orally
  Interventions: Dietary Supplement: omega-3
- placebo group (Placebo Comparator): A single dose of 4.0g corn oil was given orally
  Interventions: Dietary Supplement: placebo
- healthy control group (No Intervention): no intervention. assessement of cognitive performance twice.

INTERVENTIONS:
Dietary Supplement: omega-3 — supplement in the market
  Arms: high omega-3 group; low omega-3 group
Dietary Supplement: placebo — corn oil
  Arms: placebo group

SUMMARY:
Depression is a serious mental illness, with persistent depression and loss of interest as the main clinical manifestations, and causes varying degrees of cognitive impairment, further leading to impaired social function, and even lead to suicidal behavior. Previous studies on the antidepressant effects of Omega-3 mainly focused on chronic effects, and there was a lack of corresponding rapid response clinical studies. Because of the nature of Omega-3 health products, no clinical adverse effects have been reported. We have previously shown that Omega-3 can produce antidepressant and cognitive improvement effects. This study will carry out different doses (low dose and high dose) and single active ingredient (EPA alone) to observe the antidepressant and cognitive improvement effects of Omega-3 in clinical patients with major depression. The antidepressant effect and cognitive improvement effect of Omega-3 will be further verified to provide evidence for future clinical application.

ELIGIBILITY:
Inclusion Criteria:

* current moderate to severe depressive episode (DSM-5)
* HAMD-17>16
* 18≤Age≤45
* Never use of fluoxetine and no use of any antipsychotic and antidepressant drugs and mood stablizer at least 8 weeks
* Current physical or laboratory tests show good health
* negative usrine drug tests
* voluntray to sign the consent form

Exclusion Criteria:

* treat-resistant depressive disorder
* other axis I/II dignoses
* MMSE≤27 recent abuse history of alcohol or drugs pregnant or breast breeding

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Estimated)
Dates: Start 2022-12-15 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
depressive symptom | 40 minutes
  Hamilton Depression Scale (HAMD)-17, more reduaction mean better outcome

SECONDARY OUTCOMES:
Cognitive performance Working memory | 4 hours
  Working memory: digit span test from the Wechsler Memory Scale-Third Edition (WMS-III)
Cognitive performance Verbal memory | 4 hours
  Verbal memory: evaluate the Logical Memory including immediate/delayed recall and recognition from the WMS-III.
Cognitive performance Visual memory | 4 hours
  Visual memory: Rey-Osterrieth Complex Figure (ROCF) task
Cognitive performance | 4 hours
  executive function: the Stroop Test and the Wisconsin Card Sorting Test (WCST). more improvement mean better outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Nanfang Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No